CLINICAL TRIAL: NCT03549871
Title: ATLAS-PPX: an Open-label, Multinational, Switching Study to Describe the Efficacy and Safety of Fitusiran Prophylaxis in Patients With Hemophilia A and B Previously Receiving Factor or Bypassing Agent Prophylaxis.
Brief Title: A Study of Fitusiran in Severe Hemophilia A and B Patients Previously Receiving Factor or Bypassing Agent Prophylaxis
Acronym: ATLAS-PPX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC15110; 2016-004087-19 (EudraCT Number); ALN-AT3SC-009 (Other: Alnylam); U1111-1217-3270 (Registry Identifier: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fitusiran (Experimental): Cohort A [inhibitor]: participants with severe hemophilia A/B and inhibitory antibodies to coagulation factor VIII (FVIII)/factor IX (FIX) previously received BPA prophylaxis. Cohort B [non-inhibitor]: participants with severe hemophilia A/B without inhibitory antibodies to FVIII/FIX previously received factor prophylaxis. Participants from both cohorts was enrolled into 6-month factor/BPA prophylaxis period and continued their pre-study, regularly scheduled prophylaxis regimen with factor/BPAs. This period could be skipped by subgroup of Cohort A (hemophilia B with inhibitors to FIX and historical annualized bleeding rate [ABR] >=20) that started directly with fitusiran. Post completing factor/BPA prophylaxis period, participants entered 7-month fitusiran treatment period (1-month onset+6-month efficacy) followed by AT follow-up/roll-over into LTE15174 (NCT03754790). Throughout study, participants could receive on-demand treatment for breakthrough BE with factor/BPAs, as appropriate.
  Interventions: Drug: Fitusiran; Drug: BPA prophylaxis; Drug: Factor (FVIII or FIX) prophylaxis

INTERVENTIONS:
Drug: Fitusiran — Pharmaceutical form: solution for injection Route of administration: subcutaneous
Drug: BPA prophylaxis — Pharmaceutical form: solution for injection Route of administration: Intravenous
Drug: Factor (FVIII or FIX) prophylaxis — Pharmaceutical form: solution for injection Route of administration: Intravenous

SUMMARY:
Primary Objective:

To characterize the frequency of bleeding episodes (BE) while receiving fitusiran treatment, relative to the frequency of bleeding episodes while receiving factor concentrate or bypassing agent (BPA) prophylaxis.

Secondary Objectives:

* To characterize the following while receiving fitusiran treatment, relative to receiving factor or BPA prophylaxis:
* the frequency of spontaneous bleeding episodes
* the frequency of joint bleeding episodes
* health related quality of life (HRQOL) in participants greater than or equal to (>=) 17 years of age
* To characterize the frequency of bleeding episodes during the onset and treatment periods in participants receiving fitusiran.
* To characterize the safety and tolerability of fitusiran.
* To characterize the annualized weight-adjusted consumption of factor/BPA while receiving fitusiran treatment, relative to receiving factor or BPA prophylaxis.

DETAILED DESCRIPTION:
The estimated total time on study, inclusive of Screening, for each participant was up to 15 months for participants who were enrolled in the extension study except for participants in the subgroup of Cohort A, for whom it was up to 9 months. The estimated total time on study was up to 21 months (up to 15 months in participants in the subgroup of Cohort A) in participants who did not enroll in the extension study due to the requirement for an additional up to 6 months of follow-up for monitoring of antithrombin (AT) levels.

ELIGIBILITY:
Inclusion Criteria:

* Males, >=12 years of age.
* Severe hemophilia A or B (as evidenced by a central laboratory measurement at screening or documented medical record evidence of FVIII less than (<) 1 percent (%) or FIX level less than or equal to (<=) 2%).
* A minimum of 2 bleeding episodes required BPA treatment within the last 6 months prior to screening for participants with inhibitory antibodies to factor VIII or factor IX (Cohort A). A minimum of 1 bleeding episode required factor treatment within the last 12 months prior to screening for participants without inhibitory antibodies to factor VIII or factor IX (Cohort B).
* Met either the definition of inhibitor or non-inhibitor participant as below:
* Inhibitor: Use of BPAs for prophylaxis and for any bleeding episodes for at least the last 6 months prior to screening, and met one of the following Nijmegen-modified Bethesda assay results criteria:
* Inhibitor titer of >=0.6 Bethesda Unit per milliliter (BU/mL) at screening, or
* Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of 2 consecutive titers >=0.6 BU/mL, or
* Inhibitor titer of <0.6 BU/mL at screening with medical record evidence of anamnestic response
* The subgroup of participants in Cohort A participants might additionally meet the following criteria to be eligible to start treatment with fitusiran directly after the screening period:

  * Hemophilia B with inhibitory antibody to Factor IX as defined above
  * Not responding adequately to BPA treatment (historical ABR >=20) prior to enrollment
  * In the opinion of the Investigator, with approval of Sponsor Medical Monitor, 6-month BPA prophylaxis period should be omitted.
* Non-inhibitor: Use of factor concentrates for prophylaxis and for any bleeding episodes for at least the last 6 months prior to screening, and met each of the following criterion:
* Nijmegen-modified Bethesda assay inhibitor titer of <0.6 BU/mL at screening and
* No use of BPAs to treat bleeding episodes for at least the last 6 months prior to screening and
* No history of immune tolerance induction therapy within the past 3 years prior to screening.
* Documented prophylactic treatment with factor concentrates or BPAs for the treatment of hemophilia A or B for at least 6 months prior to screening.
* Adherent to the prescribed prophylactic therapy for at least 6 months prior to screening per Investigator assessment.
* Willed and complied with the study requirements and to provide written informed consent and assent.

Exclusion Criteria:

* Known co-existing bleeding disorders other than hemophilia A or B.
* AT activity <60% at screening.
* Co-existing thrombophilic disorder.
* Clinically significant liver disease.
* Active Hepatitis C virus infection.
* Acute or chronic Hepatitis B virus infection.
* HIV positive with a CD4 count of <200 cells per microliter.
* History of arterial or venous thromboembolism.
* Inadequate renal function.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or N-Acetylgalactosamine (GalNAc).
* History of intolerance to subcutaneous injection(s).
* Any other conditions or comorbidities that made the participant unsuitable for enrollment or could interfere with participation in or completion of the study, per Investigator judgment.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (35):
- Investigational Site Number 0139, Los Angeles, California, United States
- Investigational Site Number 6104, Prahran, Australia
- Investigational Site Number 8604, Beijing, China
- Investigational Site Number 4501, Copenhagen, Denmark
- Investigational Site Number 3303, Lyon, France
- Investigational Site Number 5301, Crumlin, Ireland
- Investigational Site Number 9701, Ramat Gan, Israel
- Investigational Site Number 3902, Milan, Italy
- Japan (4):
  - Investigational Site Number 8101, Nagoya
  - Investigational Site Number 8102, Nishinomiya
  - Investigational Site Number 8104, Saitama
  - Investigational Site Number 8109, Tokyo
- Malaysia (3):
  - Investigational Site Number 6004, Ampang
  - Investigational Site Number 6002, Johor Bahru
  - Investigational Site Number 6003, Kota Kinabalu
- Investigational Site Number 5201, San Pablo, Mexico
- South Korea (3):
  - Investigational Site Number 8201, Busan
  - Investigational Site Number 8202, Daejeon
  - Investigational Site Number 8204, Seoul
- Turkey (Türkiye) (10):
  - Investigational Site Number 9002, Adana
  - Investigational Site Number 9001, Ankara
  - Investigational Site Number 9004, Antalya
  - Investigational Site Number 9008, Gaziantep
  - Investigational Site Number 9005, Istanbul
  - Investigational Site Number 9010, Izmir
  - Investigational Site Number 9003, Izmir
  - Investigational Site Number 9009, Kayseri
  - Investigational Site Number 9006, Samsun
  - Investigational site number 9013, Van
- Ukraine (2):
  - Investigational Site Number 8003, Kyiv
  - Investigational Site Number 8002, Lviv
- United Kingdom (4):
  - Investigational Site Number 4402, Glasgow
  - Investigational Site Number 4407, London
  - Investigational Site Number 4403, London
  - Investigational Site Number 4401, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kenet G, Nolan B, Zulfikar B, Antmen B, Kampmann P, Matsushita T, You CW, Vilchevska K, Bagot CN, Sharif A, Peyvandi F, Young G, Negrier C, Chi J, Kittner B, Sussebach C, Shammas F, Mei B, Andersson S, Kavakli K. Fitusiran prophylaxis in people with hemophilia A or B who switched from prior BPA/CFC prophylaxis: the ATLAS-PPX trial. Blood. 2024 May 30;143(22):2256-2269. doi: 10.1182/blood.2023021864. PMID 38452197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 35 active sites in 15 countries. Total of 99 participants were screened from 25 July 2018 to 19 March 2021, of which 19 were screen failure due to not meeting eligibility criteria. Study had 2 main periods: 6-month factor/bypassing agent (BPA) prophylaxis period & 7-month fitusiran treatment period (1-month onset and 6-month fitusiran efficacy period).
Pre-assignment Details: Subgroup of Cohort A: Participants with hemophilia B with inhibitors and inadequate response to BPA treatment (historical annualized bleeding rate [ABR] greater than or equal to [>=] 20) prior to enrollment did not participate in 6-month prophylaxis period and they entered directly into fitusiran treatment period.
Groups:
- Cohort A: Inhibitor: Participants with hemophilia A or B and inhibitory antibodies to coagulation factor VIII (FVIII) or coagulation factor IX (FIX) and who were receiving BPA prophylaxis were enrolled in the study and entered into 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with BPAs (twice weekly [activated prothrombin complex concentrates {aPCC}] or every other day [recombinant factor VIIa {rFVIIa}]). This period was skipped by a subgroup of Cohort A (hemophilia B with inhibitors and historical ABR >= 20) and they entered directly in to fitusiran treatment period. Post completion of BPA prophylaxis period, participants entered 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 milligrams (mg) once monthly (QM) as subcutaneous (SC) injection for 7 months until the sponsor initiated a voluntary dose pause. After dose pause and protocol amendment, the fitusiran dose was changed to 50 mg once every other month (Q2M) as SC injection. Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. Throughout study, participants in fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs, as appropriate.
- Cohort B: Non-inhibitor: Participants with hemophilia A or B, without inhibitory antibodies to FVIII or FIX who were receiving factor prophylaxis were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with factor concentrates (twice weekly [standard half-life FVIII], once weekly [extended half-life FVIII; standard half-life FIX], and once biweekly [extended half-life FIX]). Post completion of factor prophylaxis period, participants entered in to 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until the sponsor initiated a voluntary dose pause. Participants could continue to receive their factor prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with factor, as appropriate.
Period: Factor/BPA Prophylaxis: Day -168 to -1
Arm/Group | Cohort A: Inhibitor | Cohort B: Non-inhibitor
Started (Enrolled) | 30 | 50
Started Directly With Fitusiran | 2 | 0
Started With Factor or BPA Prophylaxis | 28 | 50
Completed | 23 | 46
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Parent withdrew consent | 1 | 0
Not completed — Switched to treatment not per protocol | 4 | 0
Not completed — Related to Coronavrus Disease 2019 | 1 | 0
Not completed — Did not meet trial eligibility | 0 | 2
Period: Fitusiran Treatment: Day 1 to Day 190
Arm/Group | Cohort A: Inhibitor | Cohort B: Non-inhibitor
Started | 23 | 46
Received 80mg QM & Part of Safety Analysis Set 1 (SAS 1) | 21 | 46
Received 50 mg Q2M & Part of Safety Analysis Set 2 (SAS 2) | 2 (Participants received fitusiran 50mg Q2M dosing regimen after dose pause and amended protocol 5, dated 25-Nov-2020. They were considered as safety analysis set 2 (SAS 2) and were subjected only to safety analysis and not to main efficacy analysis (Efficacy Set 1).) | 0
Efficacy Analysis Set 1 (EAS 1) | 19 | 46
Efficacy Analysis Set 2 (EAS 2) | 2 (Efficacy Analysis Set 2 (EAS 2) included all participants in the SAS 2 who received BPA prophylaxis and fitusiran 50 mg Q2M after dose pause, protocol amendment 5 (dated 25-Nov-2020) and dose resumption.) | 0
Completed | 17 | 37
Not Completed | 6 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — More than 1 antithrombin (AT) measurement less than 15% | 1 | 0
Not completed — Study drug on hold | 4 | 5
Not completed — Participant's decision | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all completed participants from BPA/factor prophylaxis period + 2 participants from Cohort A subgroup who directly enrolled to fitusiran treatment period.
Groups:
- Cohort A: Inhibitor: Participants with hemophilia A or B and inhibitory antibodies to FVIII or FIX and who were receiving BPA prophylaxis were enrolled in the study and entered into 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with BPAs (twice weekly [aPCC] or every other day [rFVIIa]). This period was skipped by a subgroup of Cohort A (hemophilia B with inhibitors and historical ABR >= 20) and they entered directly in to fitusiran treatment period. Post completion of BPA prophylaxis period, participants entered 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection for 7 months until the sponsor initiated a voluntary dose pause. After dose pause and protocol amendment, the fitusiran dose was changed to 50 mg Q2M as SC injection. Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. Throughout the study, participants in fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs, as appropriate.
Arm/Group | Cohort A: Inhibitor | Cohort B: Non-inhibitor | Total Title
Number analyzed (Participants) | 23 | 46 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (15.9) | 23.5 (7.3) | 24.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 46 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 17 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 27 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Estimated Annualized Bleeding Rate (ABR)
Description: Bleeding episodes (BE): any occurrence of hemorrhage might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location occurred within 72 hours of last injection used to treat BE at that location was considered part of original BE and counted as 1 BE towards ABR. Bleeding began after 72 hours of last injection at that location was considered as a new event. ABR = total number of qualifying BE/total number of days in the respective period*365.25. Estimated data were derived by using repeated measures negative binomial (NB) regression model.
Time Frame: Factor/BPA prophylaxis period: Day -168 to Day -1 or up to last day of bleeding follow up (any day up to Day -1); 6-month fitusiran efficacy period: Day 29 to Day 190 or up to last day of bleeding follow up (any day up to Day 190), whichever was earliest
Population: Analysis was performed on efficacy analysis set 1 (EAS1) which included participants who received factor/BPA prophylaxis and any dose of fitusiran before dose resumption. Data collection and analysis of combined population of Cohort A and B for each period was planned and performed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Groups:
- Overall Factor/BPA Prophylaxis Period: All participants, whether with inhibitory antibodies (Cohort A) or without inhibitory antibodies (Cohort B) to FVIII or FIX and who were receiving BPA or factor prophylaxis were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study regularly scheduled prophylaxis regimen with BPAs (twice weekly [aPCC] or every other day [rFVIIa]) or factors (twice weekly [standard half-life FVIII], once weekly [extended half-life FVIII; standard half-life FIX], and once biweekly [extended half-life FIX]) in 6-month factor or BPA prophylaxis period. This period was skipped by a subgroup of Cohort A which included participants with hemophilia B with inhibitory antibodies to FIX and who had not responded adequately to BPA prophylaxis prior to study entry (historical ABR >=20).
- Overall Fitusiran 80 mg Efficacy Period: All participants who received fitusiran 80 mg QM as SC injection (either in Cohort A or Cohort B) until sponsor initiated a voluntary dose pause during fitusiran efficacy period (i.e., from Day 29 to Day 190 of fitusiran treatment period) and were considered for efficacy analysis during fitusiran efficacy period.
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 7.482 [5.520 to 10.141] | 2.908 [1.727 to 4.898]
Statistical Analysis 1: Comparison: Overall Factor/BPA Prophylaxis Period vs Overall Fitusiran 80 mg Efficacy Period; Analyzed using repeated measures NB model with fixed effect of treatment period (fitusiran efficacy period or factor/BPA prophylaxis period) and robust sandwich covariance matrix was constructed to account for within participant dependence, logarithm of duration (in years) that each participant spends in each study period matching BE data being analyzed as an offset variable; Test type: Superiority; p = 0.0008, Repeated measures NB regression model — The threshold for significance was <0.05; ABR ratio = 0.389, 95% CI 2-sided [0.224 to 0.675]

2. Primary Outcome: Observed Annualized Bleeding Rate (ABR)
Description: A bleeding episode (BE): any occurrence of hemorrhage might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered a part of original BE and counted as 1 BE towards ABR. Any bleeding that began after 72 hours of last injection at that location was considered as a new event. ABR = total number of qualifying BE/number of days in the respective period *365.25.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS1 population. Data collection and analysis of combined population of Cohort A and B for each period was planned and performed for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 7.56 (9.49) | 3.19 (7.75)

3. Secondary Outcome: Estimated Annualized Spontaneous Bleeding Rate
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA infusion. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered part of original BE and counted as 1 BE towards ABR. Bleeding began after 72 hours of last injection at that location was considered as a new event. Spontaneous BE: BE occurrence for no apparent/known reason, particularly into joints, muscles, and soft tissues. ABR = total number of qualifying BE/number of days in respective period *365.25. Estimated data was derived using repeated measures NB regression model.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS 1 population. Data collection and analysis of combined population of Cohort A and B for each period was planned and performed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 5.002 [3.424 to 7.305] | 2.222 [1.190 to 4.152]
Statistical Analysis 1: Comparison: Overall Factor/BPA Prophylaxis Period vs Overall Fitusiran 80 mg Efficacy Period; Test type: Superiority; ABR ratio = 0.444, 95% CI 2-sided [0.234 to 0.842]

4. Secondary Outcome: Observed Annualized Spontaneous Bleeding Rate
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered part of original BE and was counted as 1 BE towards ABR. Bleeding began after 72 hours from last injection at that location was considered as a new event. Spontaneous BE: bleeding event occurred for no apparent or known reason, particularly into joints, muscles and soft tissues. ABR = total number of qualifying BE/number of days in respective period *365.25.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 5.09 (7.93) | 2.51 (7.33)

5. Secondary Outcome: Estimated Annualized Joint Bleeding Rate
Description: BE: any hemorrhage that required administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection to treat BE at that location was considered part of original BE; counted as 1 BE towards ABR. Bleeding after 72 hours from last injection at that location was considered as a new event. Joint BE: characterized by unusual sensation in joint ("aura") + increasing swelling/warmth over joint skin, increasing pain/progressive loss of range of motion/difficulty in limb use compared to Baseline. ABR = total number of qualifying BE/number of days in respective period *365.25. Estimated data were derived by using repeated measures NB regression model.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 5.282 [3.647 to 7.651] | 2.564 [1.440 to 4.566]
Statistical Analysis 1: Comparison: Overall Factor/BPA Prophylaxis Period vs Overall Fitusiran 80 mg Efficacy Period; Test type: Superiority; ABR ratio = 0.485, 95% CI 2-sided [0.259 to 0.910]

6. Secondary Outcome: Observed Annualized Joint Bleeding Rate
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered part of original BE and counted as 1 BE towards ABR. Bleeding began after 72 hours from last injection at that location was considered as a new event. Joint BE: characterized by unusual sensation in joint (aura) increasing swelling/warmth over joint skin, increasing pain or progressive loss of range of motion/difficulty in limb use compared to Baseline. ABR = total number of joint BE/number of days in respective period*365.25.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Efficacy Period
Number analyzed (Participants) | 65 | 65
episodes per participant per year | 5.35 (8.19) | 2.82 (7.54)

7. Secondary Outcome: Change in Haemophilia Quality of Life Questionnaire for Adults (Haem-A-QOL) Physical Health Score in the Fitusiran Treatment Period and the Factor or BPA Prophylaxis Period
Description: Haem-A-QoL: participant-reported questionnaire for adults aged >=17 years with hemophilia and comprised of 46 items covering 10 domains. Physical health domain (PHD) is assessed with 5 items rated on 5-point Likert scale: never, rarely, sometimes, often or all the time. Raw score for PHD were transformed to scale ranged from 0 to 100, where lower scores = better physical health. Least square (LS) mean and 95% confidence interval (CI) by mixed model for repeated measure (MMRM) analysis with robust sandwich covariance matrix: change from Month -6 to Day 1 and to Month 7 as response variable; period (factor/BPA prophylaxis & fitusiran treatment) & Baseline score (Month -6) as fixed effects.
Time Frame: Month -6 of Factor or BPA prophylaxis period (Baseline), Day 1 (Month 1) and Month 7 of fitusiran treatment period
Population: Analysis was performed on EAS 1 population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data collection and analysis of combined population of Cohort A and B for each period was planned and performed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Overall Fitusiran 80 mg Treatment Period: All participants who received fitusiran 80 mg QM as SC injection (either in Cohort A or Cohort B) until sponsor initiated a voluntary dose pause during fitusiran treatment period (i.e., 1-month onset period + 6-month efficacy period) and were considered for efficacy analysis during fitusiran treatment period.
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Treatment Period
Number analyzed (Participants) | 48 | 48
score on a scale | -6.00 [-10.19 to -1.81] | -9.60 [-15.35 to -3.84]

8. Secondary Outcome: Change in Haemophilia Quality of Life Questionnaire for Adults Total Score in the Fitusiran Treatment Period and the Factor or BPA Prophylaxis Period
Description: Haem-A-QoL: questionnaire for adults aged >= 17 years with hemophilia; and comprised of 46 items covering 10 domains: physical health, feelings, view of yourself, sports and leisure, work and school, dealing with hemophilia, treatment, future, family planning, partnership and sexuality. Items were rated on 5-point Likert scale: never, rarely, sometimes, often or all time. Domain raw score was transformed to scale ranged from 0 to 100, where lower scores=better health. LS mean & 95% CI by MMRM analysis with robust sandwich covariance matrix: change from Month -6 to Day 1 and to Month 7 as response variable; period (factor/BPA prophylaxis & fitusiran treatment) & Baseline score (Month -6) as fixed effects.
Time Frame: Month -6 of Factor or BPA prophylaxis period (Baseline), Day 1 (Month 1) and Month 7 of fitusiran treatment period
Population: Analysis was performed on EAS1 population. Here, 'overall number of participants analyzed = participants with available data for this outcome measure. Data collection and analysis of combined population of Cohort A and B for each period was planned and performed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Overall Factor/BPA Prophylaxis Period | Overall Fitusiran 80 mg Treatment Period
Number analyzed (Participants) | 48 | 48
score on a scale | -3.07 [-5.56 to -0.58] | -7.62 [-10.26 to -4.98]

9. Secondary Outcome: Estimated Annualized Bleeding Rate in the Fitusiran Onset Period
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered part of original BE and was counted as 1 BE towards ABR. Bleeding began after 72 hours from last injection at that location was considered as new event. Estimated ABR and 95% CI was derived by using repeated measures NB regression model with logarithm of duration (years) that each participant spends in 1-Month fitusiran onset period matching BE data being analyzed as offset variable. ABR = total number of qualifying BE/number of days in respective period *365.25.
Time Frame: Day 1 up to Day 28 or up to the last day of bleeding follow up (any day up to Day 28), whichever was earliest
Population: Analysis was performed on EAS 1 population. Data collection and analysis of combined population of Cohort A and B for fitusiran 1-month onset period was planned and performed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Groups:
- Overall Fitusiran 80 mg 1-Month Onset Period: All participants who received fitusiran 80 mg QM as SC injection (either in Cohort A or Cohort B) until sponsor initiated a voluntary dose pause during fitusiran 1-month onset period and were considered for the efficacy analysis during fitusiran 1-month onset period.
Arm/Group | Overall Fitusiran 80 mg 1-Month Onset Period
Number analyzed (Participants) | 65
episodes per participant per year | 5.419 [3.716 to 7.901]

10. Secondary Outcome: Observed Annualized Bleeding Rate in the Fitusiran Onset Period
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA. BE start time: time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered a part of original BE and was counted as one BE towards ABR. Bleeding began after 72 hours from last injection at that location was considered as a new event. ABR= total number of qualifying BE/number of days in the 1-month onset period *365.25. Analysis was based on on-treatment strategy which included all treated bleeding events in 1-month onset period and excluded any bleeding events in period of intercurrent events.
Time Frame: Day 1 up to Day 28 or up to the last day of bleeding follow up (any day up to Day 28), whichever was earliest
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Overall Fitusiran 80 mg 1-Month Onset Period
Number analyzed (Participants) | 65
episodes per participant per year | 5.42 (8.28)

11. Secondary Outcome: Estimated Annualized Bleeding Rate in the Fitusiran Treatment Period
Description: BE: defined as any occurrence of hemorrhage that might require administration of factor/BPA. BE start time was time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered a part of original BE and counted as one BE towards ABR. Bleeding began after 72 hours from last injection at that location was considered as new event. Analysis was based on on-treatment strategy which included all treated bleeding events in fitusiran period and excluded any bleeding events in the period of intercurrent events. ABR = total number of qualifying BE/number of days in respective period *365.25.
Time Frame: From Day 1 up to Day 190
Population: Analysis was performed on EAS 1 population. Data collection and analysis of combined population of Cohort A and B for fitusiran treatment period was planned and performed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: episodes per participant per year
Arm/Group | Overall Fitusiran 80 mg Treatment Period
Number analyzed (Participants) | 65
episodes per participant per year | 3.317 [2.111 to 5.211]

12. Secondary Outcome: Observed Annualized Bleeding Rate in the Fitusiran Treatment Period
Description: BE: any occurrence of hemorrhage that might require administration of factor/BPA. BE start time was time at which 1st BE symptoms develop; bleeding/any symptoms at same location that occurred within 72 hours of last injection used to treat BE at that location was considered a part of original bleeding event and was counted as one BE towards ABR. Any bleeding that began after 72 hours from last injection at that location was considered as a new event. ABR= total number of qualifying BE/number of days in treatment period *365.25. Analysis was based on on-treatment strategy which included all treated bleeding events in fitusiran period and excluded any bleeding events in period of intercurrent events.
Time Frame: from Day 1 up to Day 190
Population: Analysis was performed on EAS1 population. Data collection and analysis of combined population of Cohort A and B for fitusiran treatment period was planned and performed for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes per participant per year
Arm/Group | Overall Fitusiran 80 mg Treatment Period
Number analyzed (Participants) | 65
episodes per participant per year | 3.48 (6.98)

13. Secondary Outcome: Cohort A: Annualized Weight-adjusted Consumption of BPA (Activated Prothrombin Complex Concentrates)
Description: Annualized weight-adjusted BPA consumption was calculated for each participant during prophylaxis period as: [Sum of BPA dose per body weight received during corresponding period/number of days in corresponding period]*365.25. In this outcome measure, data of annualized weight-adjusted consumption of BPA agent: aPCC (unit per kilogram [U/kg]) were reported.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS 1 population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Combined data of annualized weight-adjusted BPA consumption (U/kg) for both treated bleeds and prophylaxis purpose were reported in this outcome measure.
Measure: Mean (Standard Deviation); unit: U/kg per participant per year
Groups:
- BPA Prophylaxis: Cohort: A Inhibitor: Participants with hemophilia A or B, with inhibitory antibodies to FVIII or FIX and who were receiving BPA prophylaxis were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with BPAs ((twice weekly [aPCC] or every other day [rFVIIa]). This period was skipped by a subgroup of Cohort A which included participants with hemophilia B with inhibitory antibodies to FIX who had not responded adequately to BPA prophylaxis prior to study entry (historical ABR >=20).
- Fitusiran 80 mg Prophylaxis: Cohort A: Inhibitor: Post completion of BPA prophylaxis period, participants entered into the 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until the sponsor initiated a voluntary dose pause (up to maximum of 7 months). Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. A subgroup of Cohort A (hemophilia B participants with inhibitory antibodies to Factor IX who were not responding adequately to BPA prophylaxis prior to study entry: historical ABR >=20) entered directly into fitusiran treatment period. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs, as appropriate.
Arm/Group | BPA Prophylaxis: Cohort: A Inhibitor | Fitusiran 80 mg Prophylaxis: Cohort A: Inhibitor
Number analyzed (Participants) | 15 | 15
U/kg per participant per year | 7912.7 (5507.6) | 39.7 (87.0)

14. Secondary Outcome: Cohort A: Annualized Weight-adjusted Consumption of BPA (Recombinant Factor VIIa)
Description: Annualized weight-adjusted BPA consumption was calculated for each participant during prophylaxis period as: (Sum of BPA dose per body weight received during corresponding period/number of days in corresponding period)*365.25. In this outcome measure, data of annualized weight-adjusted consumption of BPA agents: rFVIIa (unit: micrograms per kg [mcg/kg]) were reported. Combined data of annualized weight-adjusted BPA consumption (mcg/kg) for both treated bleeds and prophylaxis purpose were reported in this outcome measure.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS 1 population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Combined data of annualized weight-adjusted BPA consumption (mcg/kg) for both treated bleeds and prophylaxis purpose were reported in this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/kg per participant per year
Groups:
- BPA Prophylaxis: Cohort: A Inhibitor: Participants with hemophilia A or B, with inhibitory antibodies to FVIII or FIX and who were receiving BPA prophylaxis were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with BPAs (twice weekly [aPCC] or every other day [rFVIIa]). This period was skipped by a subgroup of Cohort A which included participants with hemophilia B with inhibitory antibodies to FIX who had not responded adequately to BPA prophylaxis prior to study entry (historical ABR >=20).
- Fitusiran 80 mg Prophylaxis: Cohort A: Inhibitor: Post completion of BPA prophylaxis period, participants entered into the 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until the sponsor initiated a voluntary dose pause (up to maximum of 7 months). Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. A subgroup of Cohort A (hemophilia B participants with inhibitory antibodies to FIX who were not responding adequately to BPA prophylaxis prior to study entry: historical ABR >=20) entered directly into fitusiran treatment period. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs, as appropriate.
Arm/Group | BPA Prophylaxis: Cohort: A Inhibitor | Fitusiran 80 mg Prophylaxis: Cohort A: Inhibitor
Number analyzed (Participants) | 7 | 7
mcg/kg per participant per year | 18895.8 (14081.9) | 168.8 (290.8)

15. Secondary Outcome: Cohort B: Annualized Weight-adjusted Consumption of Factor
Description: Annualized weight-adjusted BPA consumption was calculated for each participant during prophylaxis period as: (Sum of BPA dose per body weight received during corresponding period/number of days in corresponding period)*365.25. In this outcome measure, data of annualized weight-adjusted consumption of BPA agents: FVIII and FIX (unit: international Units [IU] per kg [IU/kg]) were reported.
Time Frame: as for outcome 1
Population: Analysis was performed on EAS 1 population. Here, 'number analyzed' = participants with available data for each specified category. Combined data of annualized weight-adjusted factor consumption (IU/kg) for both treated bleeds and prophylaxis purpose were reported in this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/kg per participant per year
Groups:
- Factor Prophylaxis: Cohort B: Non-inhibitor: Participants with hemophilia A or B, without inhibitory antibodies to FVIII or FIX who were receiving factor prophylaxis were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with factor concentrates (twice weekly [standard half-life FVIII], once weekly [extended half-life FVIII; standard half-life FIX], and once biweekly [extended half-life FIX]).
- Fitusiran 80 mg Prophylaxis: Cohort B: Non-inhibitor: Post completion of factor prophylaxis period, participants entered in to 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until the sponsor initiated a voluntary dose pause (up to maximum of 7 months). Participants could continue to receive their factor prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with factor, as appropriate.
Arm/Group | Factor Prophylaxis: Cohort B: Non-inhibitor | Fitusiran 80 mg Prophylaxis: Cohort B: Non-inhibitor
Number analyzed (Participants) | 46 | 46
IU/kg per participant per year
  FVIII: number analyzed (Participants) | 36 | 36
  FVIII | 3396.9 (1144.5) | 60.7 (148.3)
  FIX: number analyzed (Participants) | 10 | 10
  FIX | 3175.5 (961.3) | 17.8 (56.1)

ADVERSE EVENTS:
Time Frame: Factor/BPA prophylaxis period: from Day -168 to Day -1; Fitusiran 80 mg QM/50 mg Q2M period: from Day 1 of fitusiran treatment period (i.e., 1 month onset+ 6 months efficacy) until AT follow up (i.e. up to 21 months)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug which did not necessarily have a causal relationship with the treatment. Safety analysis set (SAS): all participants who were enrolled and received any dose of fitusiran (80 mg, QM before dose pause; SAS 1)/(50 mg, Q2M after dose pause; SAS 2).
Groups:
- Cohort A: SAS 1 - BPA Prophylaxis; Cohort A: SAS 2 - BPA Prophylaxis: Participants with hemophilia A or B, with inhibitory antibodies to FVIII or FIX and who were receiving BPA prophylaxis were enrolled in the study and entered the 6-month BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with BPAs (twice weekly [aPCC] or every other day [rFVIIa]).
- Cohort A: SAS 1 - Fitusiran 80 mg QM: Post completion of BPA prophylaxis period, participants entered into the 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until sponsor initiated a voluntary dose pause. Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. A subgroup of Cohort A (participants with hemophilia B and inhibitory antibodies to FIX who had not responded adequately to BPA prophylaxis prior to study entry [historical ABR >=20]) entered directly into fitusiran treatment period. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs, as appropriate. Post last fitusiran dose, participants had a safety follow-up/AT activity level follow-up up to 6 months (monthly monitor until AT activity levels return to approximately 60% or per Investigator discretion).
- Cohort B: SAS 1 - Factor Prophylaxis: Participants with hemophilia A or B, without inhibitory antibodies to FVIII or FIX and who were receiving factor prophylaxis were enrolled in the study and entered the 6-month BPA prophylaxis period in this study and continued their pre-study, regularly scheduled prophylaxis regimen with factor concentrates (twice weekly [standard half-life FVIII), once weekly [extended half-life FVIII; standard half-life FIX], and once biweekly [extended half-life FIX]).
- Cohort B: SAS 1 - Fitusiran 80 mg QM: Post completion of Factor prophylaxis period, participants entered into the 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 80 mg QM as SC injection until sponsor initiated a voluntary dose pause (up to maximum of 7 months). Participants could continue to receive BPA prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with factor, as appropriate. Post last fitusiran dose, participants had a safety follow-up/AT activity level follow-up up to 6 months (monthly monitor until AT activity levels return to approximately 60% or per Investigator discretion).
- Overall: SAS 1 - Factor/BPA Prophylaxis: All participants whether with inhibitory antibodies (Cohort A) or without inhibitory antibodies (Cohort B) to FVIII or FIX and who were receiving BPA or factor prophylaxis, respectively, were enrolled in the study and entered the 6-month factor or BPA prophylaxis period in this study and continued their pre-study regularly scheduled prophylaxis regimen with BPAs (twice weekly [aPCC] or every other day [rFVIIa]) or factors (twice weekly [standard half-life FVIII), once weekly [extended half-life FVIII; standard half-life FIX], and once biweekly [extended half-life FIX]) in 6-month factor or BPA prophylaxis period. This period was skipped by a subgroup of Cohort A which included participants with hemophilia B with inhibitory antibodies to FIX and who had not responded adequately to BPA prophylaxis prior to study entry (historical ABR >=20).
- Overall: SAS 1 - Fitusiran 80 mg QM: Post completion of BPA prophylaxis period, all participants who received fitusiran 80 mg QM as SC injection (either in Cohort A or Cohort B) until sponsor initiated a voluntary dose pause (up to maximum of 7 months). Participants could continue to receive BPA/factor prophylaxis for up to 7 days after start of fitusiran treatment on Day 1. A subgroup of Cohort A (participants with hemophilia B and inhibitory antibodies to FIX who had not responded adequately to BPA prophylaxis treatment [historical ABR >=20]) entered directly into fitusiran treatment period. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs or factors, as appropriate. Post last fitusiran dose, participants had a safety follow-up/AT activity level follow-up up to 6 months (monthly monitor until AT activity levels return to approximately 60% or per Investigator discretion).
- Cohort A: SAS 2 - Fitusiran 50 mg Q2M: Post completion of BPA prophylaxis period, participants entered into the 7-month fitusiran treatment period (1-month onset period + 6-month efficacy period) and received fitusiran 50 mg Q2M as SC injection after sponsor initiated voluntary dose pause and protocol amendment. Throughout the study, participants in the fitusiran treatment period could receive on-demand treatment for breakthrough bleeding episodes with BPAs (twice weekly [aPCC] or every other day [rFVIIa]), as appropriate. Post last fitusiran dose, participants had a safety follow-up/AT activity level follow-up up to 6 months (monthly monitor until AT activity levels return to approximately 60% or per Investigator discretion).
Arm/Group | Cohort A: SAS 1 - BPA Prophylaxis | Cohort A: SAS 1 - Fitusiran 80 mg QM | Cohort B: SAS 1 - Factor Prophylaxis | Cohort B: SAS 1 - Fitusiran 80 mg QM | Overall: SAS 1 - Factor/BPA Prophylaxis | Overall: SAS 1 - Fitusiran 80 mg QM | Cohort A: SAS 2 - BPA Prophylaxis | Cohort A: SAS 2 - Fitusiran 50 mg Q2M
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/46 | 0/46 | 0/65 | 0/67 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/19 | 5/21 | 0/46 | 4/46 | 5/65 | 9/67 | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 10/19 | 13/21 | 9/46 | 28/46 | 19/65 | 41/67 | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: SAS 1 - BPA Prophylaxis (N=19) | Cohort A: SAS 1 - Fitusiran 80 mg QM (N=21) | Cohort B: SAS 1 - Factor Prophylaxis (N=46) | Cohort B: SAS 1 - Fitusiran 80 mg QM (N=46) | Overall: SAS 1 - Factor/BPA Prophylaxis (N=65) | Overall: SAS 1 - Fitusiran 80 mg QM (N=67) | Cohort A: SAS 2 - BPA Prophylaxis (N=2) | Cohort A: SAS 2 - Fitusiran 50 mg Q2M (N=2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemophilic Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular Device Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central Venous Catheter Removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma Late Onset (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: SAS 1 - BPA Prophylaxis (N=19) | Cohort A: SAS 1 - Fitusiran 80 mg QM (N=21) | Cohort B: SAS 1 - Factor Prophylaxis (N=46) | Cohort B: SAS 1 - Fitusiran 80 mg QM (N=46) | Overall: SAS 1 - Factor/BPA Prophylaxis (N=65) | Overall: SAS 1 - Fitusiran 80 mg QM (N=67) | Cohort A: SAS 2 - BPA Prophylaxis (N=2) | Cohort A: SAS 2 - Fitusiran 50 mg Q2M (N=2)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Buttock Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (3) | 3 (3) | 0 (0) | 15 (19) | 1 (3) | 18 (22) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (3) | 0 (0) | 3 (4) | 1 (1) | 4 (7) | 0 (0) | 0 (0)
Fibrin D Dimer Increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Lymphocyte Count Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 4 (8) | 4 (5) | 5 (9) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 7 (9) | 1 (1) | 8 (10) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (4) | 4 (5) | 1 (1) | 2 (2) | 4 (5) | 6 (7) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03549871/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03549871/SAP_001.pdf